CLINICAL TRIAL: NCT01482741
Title: Understanding Patient Perspectives on the Risks of Ionizing Radiation Used for Medical Imaging
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-185
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Colon Cancer; Lung Cancer; Neuroblastoma; Testicular Cancer
Keywords: Quality of Life; Focus groups; Risks of Ionizing Radiation; Risk of medical imaging; 11-185
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Neuroblastoma; Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Pts undergoing chemotherapy for Stage IV colorectal carcinoma: Six focus groups of 7-9 participants each will be conducted for approximately 90 minutes according to the established methodology of Krueger and Casey. Focus group sessions are semi-structured group interviews in which previously chosen, open-ended questions about topics of interest are posed to participants by a trained moderator.
  Interventions: Behavioral: Focus Group Sessions
- Parents of pediatric patients stage 1-3 neuroblastoma: within the preceding 6 months. Six focus groups of 7-9 participants each will be conducted for approximately 90 minutes according to the established methodology of Krueger and Casey. Focus group sessions are semi-structured group interviews in which previously chosen, open-ended questions about topics of interest are posed to participants by a trained moderator.
  Interventions: Behavioral: Focus Group Sessions
- Women who have undergone tx for early stage breast cancer: within the preceding 6 months. Six focus groups of 7-9 participants each will be conducted for approximately 90 minutes according to the established methodology of Krueger and Casey. Focus group sessions are semi-structured group interviews in which previously chosen, open-ended questions about topics of interest are posed to participants by a trained moderator.
  Interventions: Behavioral: Focus Group Sessions
- Men undergoing surveillance imaging after tx for testicular ca: Six focus groups of 7-9 participants each will be conducted for approximately 90 minutes according to the established methodology of Krueger and Casey. Focus group sessions are semi-structured group interviews in which previously chosen, open-ended questions about topics of interest are posed to participants by a trained moderator.
  Interventions: Behavioral: Focus Group Sessions
- Men & women enrolled in the MSKCC lung ca screening program: Six focus groups of 7-9 participants each will be conducted for approximately 90 minutes according to the established methodology of Krueger and Casey. Focus group sessions are semi-structured group interviews in which previously chosen, open-ended questions about topics of interest are posed to participants by a trained moderator.
  Interventions: Behavioral: Focus Group Sessions
- Men and women enrolled in the thoracic survivorship: Six focus groups of 7-9 participants each will be conducted for approximately 90 minutes according to the established methodology of Krueger and Casey. Focus group sessions are semi-structured group interviews in which previously chosen, open-ended questions about topics of interest are posed to participants by a trained moderator.
  Interventions: Behavioral: Focus Group Sessions

INTERVENTIONS:
Behavioral: Focus Group Sessions — Participants will complete a pre-focus group demographic questionnaire. Focus group participants will be asked to report the following: current age; gender; race/ethnicity; income; highest education attained; occupation; and cancer stage if participant has a cancer history. Participants who are parents of pediatric patients will also report their child's current age, gender, and cancer stage. Ten questions will be developed by the investigators and posed to each group by the moderator to solicit the desired information. The objective for the focus groups will be to systematically explore three domains: 1) what participants know about radiation as it relates to medical imaging; 2) how what they know or believe about radiation shapes their attitudes about it; 3) and participant perceptions regarding the availability and adequacy of their sources, including risk-benefit communication with health care providers
  Groups: Pts undergoing chemotherapy for Stage IV colorectal carcinoma
Behavioral: Focus Group Sessions — Participants will complete a pre-focus group demographic questionnaire. Focus group participants will be asked to report the following: current age; gender; race/ethnicity; income; highest education attained; occupation; and cancer stage if participant has a cancer history. Participants who are parents of pediatric patients will also report their child's current age, gender, and cancer stage. Ten questions will be developed by the investigators and posed to each group by the moderator to solicit the desired information. The objective for the focus groups will be to systematically explore three domains: 1) what participants know about radiation as it relates to medical imaging; 2) how what they know or believe about radiation shapes their attitudes about it; 3) and participant perceptions regarding the availability and adequacy of their sources, including risk-benefit communication with health care providers
  Groups: Parents of pediatric patients stage 1-3 neuroblastoma
Behavioral: Focus Group Sessions — Participants will complete a pre-focus group demographic questionnaire. Focus group participants will be asked to report the following: current age; gender; race/ethnicity; income; highest education attained; occupation; and cancer stage if participant has a cancer history. Participants who are parents of pediatric patients will also report their child's current age, gender, and cancer stage. Ten questions will be developed by the investigators and posed to each group by the moderator to solicit the desired information. The objective for the focus groups will be to systematically explore three domains: 1) what participants know about radiation as it relates to medical imaging; 2) how what they know or believe about radiation shapes their attitudes about it; 3) and participant perceptions regarding the availability and adequacy of their sources, including risk-benefit communication with health care providers
  Groups: Women who have undergone tx for early stage breast cancer
Behavioral: Focus Group Sessions — Participants will complete a pre-focus group demographic questionnaire. Focus group participants will be asked to report the following: current age; gender; race/ethnicity; income; highest education attained; occupation; and cancer stage if participant has a cancer history. Participants who are parents of pediatric patients will also report their child's current age, gender, and cancer stage. Ten questions will be developed by the investigators and posed to each group by the moderator to solicit the desired information. The objective for the focus groups will be to systematically explore three domains: 1) what participants know about radiation as it relates to medical imaging; 2) how what they know or believe about radiation shapes their attitudes about it; 3) and participant perceptions regarding the availability and adequacy of their sources, including risk-benefit communication with health care providers
  Groups: Men undergoing surveillance imaging after tx for testicular ca
Behavioral: Focus Group Sessions — Participants will complete a pre-focus group demographic questionnaire. Focus group participants will be asked to report the following: current age; gender; race/ethnicity; income; highest education attained; occupation; and cancer stage if participant has a cancer history. Participants who are parents of pediatric patients will also report their child's current age, gender, and cancer stage. Ten questions will be developed by the investigators and posed to each group by the moderator to solicit the desired information. The objective for the focus groups will be to systematically explore three domains: 1) what participants know about radiation as it relates to medical imaging; 2) how what they know or believe about radiation shapes their attitudes about it; 3) and participant perceptions regarding the availability and adequacy of their sources, including risk-benefit communication with health care providers
  Groups: Men & women enrolled in the MSKCC lung ca screening program
Behavioral: Focus Group Sessions — Participants will complete a pre-focus group demographic questionnaire. Focus group participants will be asked to report the following: current age; gender; race/ethnicity; income; highest education attained; occupation; and cancer stage if participant has a cancer history. Participants who are parents of pediatric patients will also report their child's current age, gender, and cancer stage. Ten questions will be developed by the investigators and posed to each group by the moderator to solicit the desired information. The objective for the focus groups will be to systematically explore three domains: 1) what participants know about radiation as it relates to medical imaging; 2) how what they know or believe about radiation shapes their attitudes about it; 3) and participant perceptions regarding the availability and adequacy of their sources, including risk-benefit communication with health care providers
  Groups: Men and women enrolled in the thoracic survivorship

SUMMARY:
Risks from imaging-related radiation exposure have become a popular topic in the media. Because these tests are commonly applied to patients at a cancer center, it is important to understand what patients know, how they feel about what they know, where they get their information, and how satisfied they are with available risk-benefit communication on this topic.

The purpose of this study is to understand how cancer patients perceive risks and benefits of diagnostic radiation and their satisfaction with healthcare communication on this topic.

ELIGIBILITY:
Inclusion Criteria:

* English-language fluent
* 18 years of age, or older
* Provide informed consent
* Group 1: Patients undergoing chemotherapy for Stage IV colorectal carcinoma.
* Group 2: Parents of pediatric patients who have undergone treatment for stage 1-3 neuroblastoma.
* Group 3: Women who have undergone treatment for early stage breast cancer within the preceding 6 months.
* Group 4: Men undergoing surveillance imaging after treatment for testicular cancer.
* Group 5: Patients currently or previously enrolled in the MSKCC lung cancer screening program.
* Group 6: Patients enrolled in or eligible for the thoracic survivorship program.

Exclusion Criteria:

* Participants who don't speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinical practices at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
characterize participant knowledge, attitudes | 2 years
  about imaging radiation, information sources, and satisfaction with risk-benefit communication.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Thornton, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/